CLINICAL TRIAL: NCT05381883
Title: Mental Health of Professionals of the Silver Economy of New Aquitaine : Online Survey of Accommodation Establishments for Old People and Home Assistance Establishments
Acronym: SILVER NA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A01953-38
Record Dates: First submitted 2022-05-06; First posted 2022-05-19 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: COVID-19 Pandemic; Professional Stress
Keywords: COVID-19; Health Professionals; Psychological troubles; Health institution
MeSH Terms: conditions — COVID-19; Occupational Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidemiology (Other): Participants will answer sociodemographic questions, questions about the experience of potentially traumatic lifelong events, the presence of a known psychological or medical disorder and the taking of drug treatment.
  These questionnaires will make it possible to detect the main psychological disorders (post-traumatic stress disorder, depression, panic disorder, generalized anxiety disorder), to evaluate coping strategies, the presence of professional exhaustion (burnout), the consumption of psychoactive substances and quality of life.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Participants will answer socio-demographic questions, questions about the lifetime experience of potentially traumatic events, the presence of a known psychological or medical disorder and the taking of medication, and a series of psychological assessment questionnaires.
  The questionnaires, performed outside routine care, are as follows :
  Posttraumatic stress disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders-5 Beck Depression Inventory-Fast Screen General Anxiety Disorder-7 Coping Inventory for Stressful Situations Maslach Burnout Inventory Medical Outcomes Study Short-Form
  The total time for completing the questionnaires is estimated at 20 minutes

SUMMARY:
The purpose of this study is identify the psychological impact of the coronavirus-19 pandemic on professionals in residential care facilities for old people and home help professionals in New-Aquitaine by :

1. Large-scale screening for the prevalence of mental health disorders among staff.
2. Identification of vulnerability and resilience factors.
3. Improving access to early care for affected professionals.

DETAILED DESCRIPTION:
This is a repeated cross-sectional descriptive study with two independent collection points six months apart, using socio-economic self-questionnaires and psychometric scales, which aims to measure the incidence of psychological disorders.

This study included the completion of questionnaires in a non-clinical population. This is a study aimed at describing a profile of psychological condition in adults.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 and over,
* Have given their consent to participate in the study,
* Work in an accommodation establishment for the elderly or professional home help in New Aquitaine.
* Master the French language.
* Accept online reviews
* Be a beneficiary of health insurance

Exclusion Criteria:

* Bad understanding of instructions making consent or assessment impossible
* Refusal to participate
* Be under measure of legal protection: guardianship, trusteeship or safeguard of justice

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anxiety disorders | Baseline
  The appearance of symptoms of anxiety disorders measured through the General Anxiety Disorder-7 questionnaire A total score greater than 7 should lead to the hypothesis of a generalized anxiety disorder. A total score between 5 and 9 corresponds to mild anxiety, a score of 10 to 14 corresponds to moderate anxiety and a score above 15 corresponds to severe anxiety.
Prevalence of anxiety disorders | Baseline
  The appearance of symptoms of anxiety disorders measured through the Panic Disorder Self-Report questionnaire. This questionnaire is a 24-item self-report measure designed to diagnose panic disorder based on Diagnostic and Statistical Manual-IV and Diagnostic and Statistical Manual-V criteria.
  Most of items are answered in a simple Yes/No fashion. Nevertheless, there are also some questions, for example about severity, which are answered on 5-point Likert scales. Not all of the questions have to be answered by every patient. If a panic disorder can already be excluded, the questionnaire stops.

SECONDARY OUTCOMES:
Measure the prevalence of post-traumatic stress disorder | Baseline
  Participants will answer the Posttraumatic stress disorder Checklist which is a questionnaire allowing the screening of post-traumatic stress disorder.
  Min=0 max=80 Higher score mean a worse outcome
Measure the prevalence of depressive episodes | Baseline
  Participants will answer the Beck Depression Inventory- Fast Screen which is the questionnaire for screening for major depressive disorder Min = 0 Max =21 Higher score mean a worse outcome
Measure the prevalence of depressive episodes | Baseline
  Participants will answer the Coping Inventory for Stressful Situations which is the scale assesses the 4 types of coping strategies (emotion-focused, support-focused, problem-focused, avoidance-focused ).
  There are three sub-scales :
  Task oriented min=0 max=56 Emotional oriented min=0 max =42 Avoidance oreinted min =0 max =51
Study the professional burnout syndrome | Baseline
  Participants will answer the Maslach Burnout Inventory which is the questionnaire allowing the screening of a burn-out.
  There are three sub-scales :
  Burnout score min =0 max =54 Depersonalization score / Loss of empathy min =0 max=30 For these two subscales: Higher scores mean a worse outcome Personal Achievement Score min = 0 max=48 For this subscale: Higher score mean a better outcome
Study the the quality of life at work among staff | Baseline
  Participants will answer the Medical Outcomes Study Short-Form which is the questionnaire to assess the quality of life Min=0 max=100 Higher score mean a better outcome
Study the use of psychostimulant substances (drugs, alcohol, drugs, tobacco) among the staff of accommodation facilities for old people and home help | Baseline
  The consumption of psychoactive substances will be assessed through a multiple-choice menu, allowing to tick the substances consumed by the participant during the last month. The categories of psychoactive substances are: anxiolytics and sedatives (eg benzodiazepines, hypnotics etc), psycho-stimulants (eg cocaine, amphetamines, ecstasy etc), opiates and related drugs (eg codeine, heroin etc), cannabis, alcohol and tobacco. According to the items, the person will indicate for each psychoactive substance checked the level of consumption (absent, new, increasing, constant).

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Henry MARTIN, MD, Study Director — Physician
Locations (1):
- Centre Hospitalier Charles Perrens, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mohammed A, Sheikh TL, Poggensee G, Nguku P, Olayinka A, Ohuabunwo C, Eaton J. Mental health in emergency response: lessons from Ebola. Lancet Psychiatry. 2015 Nov;2(11):955-7. doi: 10.1016/S2215-0366(15)00451-4. No abstract available. PMID 26544738
- [Result] Chan AO, Huak CY. Psychological impact of the 2003 severe acute respiratory syndrome outbreak on health care workers in a medium size regional general hospital in Singapore. Occup Med (Lond). 2004 May;54(3):190-6. doi: 10.1093/occmed/kqh027. PMID 15133143
- [Result] Chua SE, Cheung V, McAlonan GM, Cheung C, Wong JW, Cheung EP, Chan MT, Wong TK, Choy KM, Chu CM, Lee PW, Tsang KW. Stress and psychological impact on SARS patients during the outbreak. Can J Psychiatry. 2004 Jun;49(6):385-90. doi: 10.1177/070674370404900607. PMID 15283533
- [Result] Csikszentmihalyi M, Larson R. Validity and reliability of the Experience-Sampling Method. J Nerv Ment Dis. 1987 Sep;175(9):526-36. doi: 10.1097/00005053-198709000-00004. PMID 3655778
- [Result] Greenberg N, Docherty M, Gnanapragasam S, Wessely S. Managing mental health challenges faced by healthcare workers during covid-19 pandemic. BMJ. 2020 Mar 26;368:m1211. doi: 10.1136/bmj.m1211. No abstract available. PMID 32217624